CLINICAL TRIAL: NCT07339995
Title: Fertility Outcomes of Ovarian Tissue Cryopreservation
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: PAED-2025-067
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ovarian tissue freezing and subsequent auto-transplantation after thawing — Removal of the ovarian tissue will be retrieved via laparoscopic surgery under general anesthesia. The ovarian cortical tissue obtained will be transferred on ice to the laboratory for cryopreservation. After medical treatment, if the patient would like to start a family but has experienced premature ovarian failure, she will have ovarian tissue auto-transplantation after thawing.

SUMMARY:
With the advancement of assisted reproductive technology, more young cancer patients can consider having children. Ovaries and testes are important reproductive organs, and drugs, diseases, chemotherapy, and radiotherapy can all damage them. Reproductive preservation technology aims to protect patients whose reproductive ability has been damaged due to gonadotoxic drug therapy. Women can preserve their reproductive ability by freezing ovarian tissue cryopreservation so that they can have children in the future. Patients who have undergone or will undergo ovarian tissue cryopreservation in Hong Kong Children's Hospital will be invited to participate in the study. Here, we aim to evaluate the outcomes after ovarian tissue cryopreservation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 0-18 years old and diagnosed with cancer
* Patients who have undergone or will undergo ovarian tissue cryopreservation in Hong Kong Children's Hospital
* For patients under 18 years old, parents/legal guardians will be asked to further sign the consent for them.

Exclusion Criteria:

* Patients unable to provide consent/assent (i.e. significant psychiatric problems/cognitive delay)
* Male patients

Ages: 0 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Patients who have undergone or will undergo ovarian tissue cryopreservation in the Hong Kong Children's Hospital will be invited to join this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2031-01-14 (Estimated); Study Completion 2032-01-14 (Estimated)

PRIMARY OUTCOMES:
Surgical complications | 15 years
  Surgical complications after ovarian tissue transplantation
Pregnancy rate | 15 years
  Pregnancy rate after ovarian tissue transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Pui Wah Jacqueline Chung, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided